CLINICAL TRIAL: NCT05773092
Title: A Phase 2 Study of Osimertinib and S-1 in Treatment Resistant EGFR Mutant NSCLC (SOS-1 Study)
Brief Title: A Phase 2 Study of Osimertinib and S-1 in Treatment Resistant EGFR Mutant NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022/2640
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: NSCLC
Keywords: EGFR mutant lung cancer; Progression on Osimertinib
MeSH Terms: interventions — S 1 (combination); osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Oral S-1 + Oral Osimertinib
  Interventions: Drug: Oral S-1 + Oral Osimertinib

INTERVENTIONS:
Drug: Oral S-1 + Oral Osimertinib — S-1 (40mg) will be given orally twice a day (daily) from Day 1 to 14 (21 day cycle), and Osimertinib (80mg) will be given orally daily continuously.

SUMMARY:
The objective of this study is to determine best overall response rate (BOR) based on radiological assessment per RECIST v1.1 to combination of S-1 and Osimertinib in treatment-resistant EGFR mutant lung cancer.

DETAILED DESCRIPTION:
A lead-in phase of 6 patients will be initiated prior to the formal phase II study. The planned sample size is 27 patients (lead-in and phase II).

The primary objective of the study is to demonstrate that S-1 fixed dose 40 mg BD is safe and effective in EGFR metastatic lung cancer resistant to Osimertinib in terms of best overall response (BOR).

The secondary objective of this study will be to further analyse the Disease Control Rate at stipulated timepoints (6,12 and 24 months), Progression-free survival, Overall Survival, and also the Toxicity by CTCAE 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed EGFR mutant NSCLC.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral CT scan, MRI, or calipers by clinical exam.
* Prior therapy: Patient with recurrent and/or metastatic EGFR mutant NSCLC, that has progressed on osimertinib as most recent line of treatment, and the primary doctor intends to continue with osimertinib treatment.
* Patients with no matched alterations (tumor or plasma) where clinical trials or approved systemic anti-cancer therapy are available, are eligible
* Patients with matched alterations on rebiopsy (tumor or plasma) who declined matching clinical trials, or approved systemic anti-cancer therapy, are eligible
* Age ≥21 years.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Patients must have adequate organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤ institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
  * creatinine ≤ institutional ULN OR glomerular filtration rate (GFR) ≥50 mL/min/1.73 m2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial provided that DDI with osimertinib has been addressed.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
* Patients with asymptomatic new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* The effects of S-1 on the developing human fetus are unknown. For this reason and because cytotoxic agents are known to be teratogenic, women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of treatment. Women must not be breastfeeding. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* Patients who are receiving any other investigational agents.
* Patients are excluded if they have symptomatic brain metastases or leptomeningeal metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to S-1.
* Concomitant medications: Patients should only be excluded from trial participation when clinically relevant known or predicted drug-drug interactions or potential overlapping toxicities will impact safety or efficacy. Please include scientific or clinically based rationale for exclusion.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations
* Pregnant women are excluded from this study because both compounds are potentially teratogenic.
* Subjects with concomitant second malignancies (except adequately treated non-melanomatous skin cancers, in situ cervical cancers, localized prostate cancer or in situ breast cancer) are excluded unless a complete remission was achieved at least 3 years prior to study entry and no additional therapy is required or anticipated to be required
* Prior organ allograft or allogeneic bone marrow transplantation
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
* Inability to comply with restrictions and prohibited activities/treatments in this study.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  The efficacy of S-1 and Osimertinib. ORR is defined as the proportion of subjects who have best objective response (BOR) of CR or PR from start of combination treatment until disease progression or death due to any cause.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with a best response of CR, PR or SD.
Progression-free survival (PFS) | Up to 3 years after end of treatment
  PFS is defined as time from study entry until objective tumour progression, or death from any cause, whichever occurs first.
Overall survival (OS) | Up to 3 years after end of treatment
  OS is defined as time from study entry to death (from any cause).

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wan-Teck Lim, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Center Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No